CLINICAL TRIAL: NCT05549739
Title: Evaluation of Respiratory Parameters and Functional Capacity in Coronary Artery Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Dilara Saklica, Principal Investigator, Hacettepe University
Other Study IDs: GO 20/298
Record Dates: First submitted 2022-09-18; First posted 2022-09-22 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease
Keywords: respiratory function test; physical functional performance; coronary artery disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: Individuals without cardiac and pulmonary disease
- Study Group: Individuals with coronary artery disease

SUMMARY:
The purpose of this study is to evaluate respiratory parameters and functional capacity in coronary artery patients.

DETAILED DESCRIPTION:
Decreased pulmonary function as measured by forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), or peak expiratory flow (PEF) has been associated with an increased risk of cardiovascular mortality and morbidity. A low MIP value may generally indicate weak muscle strength and therefore be an indicator of general poor health. Respiratory muscle weakness and decreased respiratory muscle endurance affect exercise tolerance in individuals with chronic disease, including cardiovascular disease. Studies have supported the association of grip strength with frailty, physical activity, diabetes, functional limitation, nutritional status, metabolic syndrome, and mortality.

The study will evaluate respiratory parameters and functional capacity in coronary artery patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease
* Volunteering to participate in the research

Exclusion Criteria:

* Having a musculoskeletal problem
* Having unstable cardiac disease
* Having chronic heart failure (NYHA III-IV)
* A history of acute coronary syndrome or surgical revascularization less than 3 months ago
* Having arrhythmia
* Having the last stage of kidney disease
* Having active myocarditis or pericarditis

Ages: 41 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are more than 40 years old and diagnosed with coronary artery disease.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Six-minute-step test | Day 1
  The number of steps the participant climbed up and down is recorded.
Respiratory muscle strength | Day 1
  Respiratory muscle strength will be evaluated using a mouth pressure device.
Respiratory muscle endurance | Day 1
  Respiratory muscle endurance will be evaluated using a constant load test.

SECONDARY OUTCOMES:
Pulmonary functions | Day 1
  Forced vital capacity (FVC), Forced expiratory volume at one second (FEV1), Peak expiratory flow (PEF) assessment via spirometry.
Hand grip strength | Day 1
  Hand grip strength is evaluated by a hand dynamometer.
Functional Capasity | Day 1
  The functional capacity is assessed with The Duke Activity Status Index (DASI).

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Vardar-Yagli, PhD, Study Director — Hacettepe University; Hikmet Yorgun, PhD, Study Director — Hacettepe University; Ahmet Hakan Ates, PhD, Study Chair — Hacettepe University; Dilara Saklica, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)